CLINICAL TRIAL: NCT06571071
Title: A Randomized, Double Blind, Placebo-controlled, Parallel Arm Clinical Trial of De-Stress & Chill Gummies in Reducing Stress and Anxiety, and Improving Mood in Adults
Brief Title: A Clinical Study of De-Stress & Chill Gummies in Reducing Stress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herbolab India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MHC/CT/24-25/016; CTRI/2024/07/071254 (Registry Identifier: Clinical trial registry of India)
Record Dates: First submitted 2024-08-10; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Stress; Anxiety
Keywords: stress; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, Double blind, Parallel Group, Placebo Controlled Trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- De-Stress and Chill Gummies-U001 (Experimental)
  Interventions: Other: De-Stress and Chill Gummies-U001
- De-Stress and Chill Gummies-I001 (Experimental)
  Interventions: Other: De-Stress and Chill Gummies-I001
- Placebo Gummies-001 (Placebo Comparator)
  Interventions: Other: Placebo Gummies-001

INTERVENTIONS:
Other: De-Stress and Chill Gummies-U001 — Two gummies in sequence daily after meal for 60 days
  Arms: De-Stress and Chill Gummies-U001
Other: De-Stress and Chill Gummies-I001 — Two gummies in sequence daily after meal for 60 days
  Arms: De-Stress and Chill Gummies-I001
Other: Placebo Gummies-001 — Two gummies in sequence daily after meal for 60 days
  Arms: Placebo Gummies-001

SUMMARY:
The current study focuses on clinical validation of efficacy of nutraceutical product in reduction of stress,anxiety and improving mood in adults. Adults experiencing chronic stress and anxiety often suffer from a reduced quality of life, marked by symptoms such as irritability, fatigue, and difficulty concentrating. By integrating these gummies into their daily routine, many report noticeable improvements in their emotional and mental state. These enhancements can manifest as increased energy levels, better sleep quality, and a more balanced mood, which collectively contribute to a more positive outlook on life.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-arm, comparative, multicenter, placebo-controlled, clinical trial of De-Stress and Chill Gummies in reducing stress and anxiety, and improving mood in adults.

In this study, more than 72 participants will be enrolled and randomized into one of the following groups to achieve at least 72 completers (at least 24 participants in each group): Group A: De-Stress and Chill Gummies-U001, Group B: De-Stress and Chill Gummies-I001, and Group C: Placebo Gummies-001, in a 1:1:1 ratio. The study duration is 68 days. The efficacy of the investigational products will be compared between the groups.

Concomitant diseases/medication assessment will be performed at screening.

Assessment of changes in perceived stress scale (PSS) score, LDH and creatine kinase levels, body weight and BMI, mental chatter score using 5-point scale, Hamilton Anxiety Rating Scale (HAM-A) score, COPE Questionnaire (a. Positive Subscale b. Denial Subscale) score, STAI (State-Trait Anxiety Inventory) score, visual analogue scale score- for evaluation of fatigue, nausea, palpitation, breathlessness, will be done at screening, day 30 and day 60. Assessment of changes in serum cortisol levels will be done at screening, day 15 and day 60. Assessment of changes in serotonin levels will be done at screening, day 30 and day 45. Assessment of changes in Profile of Mood State (POMS) questionnaire score (a. Total Mood Disturbance b. Depression) will be done at screening, day 15, day 30, and day 60. Assessment of modified sleep regularity and medication withdrawal questionnaire (MSRMWQ) score after stopping treatment for 1 week (day 68).

Assessment of changes in vital sign parameters will be done at baseline, Day 15, Day 30, Day 45, and Day 60. Assessment of changes in complete blood count, liver function test and kidney function test at screening and Day 60. Safety of the investigational treatment in terms of adverse events (AEs), and serious adverse events (SAEs) will be assessed at baseline, Day 15, Day 30, Day 45 and Day 60. Treatment compliance and tolerability will be assessed at Day 30 and Day 60.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 21-50 years both inclusive
2. Suffering from self-reported mild to moderate stress on the PSS scale score less than or equal to 26
3. Participants willing to participate in clinical trials and who have read understood and signed the informed consent form
4. No severe anxiety and depression i.e. Generalized anxiety disorder GAD score less than or equal to 10 and Patients' health questionnaire-9 PHQ-9 score less than or equal to 14
5. A female participant who is of reproductive potential has a negative pregnancy test and agrees to use contraception throughout the study period 6 No history of substance use disorder other than the use of nicotine and recreational use of alcohol not having used for the last 14 days and consenting not to use the same during the period of the trial

7. Willing to limit caffeine consumption while in the study.

Exclusion Criteria:

1. Inability to perform any of the assessments required for endpoint analysis
2. Shows signs of dementia, such as caused by Alzheimer's Disease, acquired immunodeficiency syndrome (AIDS), Creutzfeldt-Jakob disease (CJD), Lewy Bodies dementia (LBD), Cerebrovascular dementia (CVD), Progressive Supranuclear Palsy (PSP), multiple cerebral infarctions, or normal pressure hydrocephalus (NPH)
3. Participants currently using any nutraceutical, allopathic, or ayurvedic supplement for stress management
4. Have any other neurodegenerative diseases or seizure disorder
5. Known hypersensitivity to investigational products
6. Participants with a history of malignancy diagnosed within the past 5 years or currently diagnosed with malignancy
7. Pregnant or lactating women, as well as women of childbearing potential who are not using contraception or intending to conceive during the study
8. Sitting or resting systolic blood pressure of more than 180 mm Hg or diastolic blood pressure of more than 110 mm Hg at screening
9. Participants with a history of substance abuse, drugs, heavy use of alcohol, and/or smoking within the last 5 years
10. Serious illness or any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the participant or preclude the successful completion of the study.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Screening, day 30, day 60
  The PSS-10 is widely used for measuring psychological distress. It contains 10 questions on a five-point scale from 0 to 4. The higher the score, the greater the feeling of stress. PSS-10 Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Changes in Creatine kinase | Screening, day 30, day 60
  Blood level of Creatine kinase was measured. (U/L)
Changes in Lactate dehydrogenase(LDH) | Screening, day 30, day 60
  Blood level Lactate dehydrogenase of was measured. (U/L)
Body Mass Index (BMI) | Screening, day 30, day 60
  Body Mass Index (BMI) will be calculated using the standard formula from participants' height and weight. BMI = (Weight in Pounds / (Height in inches x Height in inches)) x 703
Mental chatter 5-point scale | Screening, day 30, day 60
  Grading will be assessed on a 5-point ordinal scale. Score assessment according to the following- 1-High mental chatter, 2-Moderate mental chatter, 3-Less but frequent mental chatter, 4-less and rare mental chatter, 5-no mental chatter
Assessment of anxiety using Hamilton Anxiety Rating Scale (HAM-A) | Screening, day 30, day 60
  Participants will be interviewed by mental health professionals using the clinically validated Hamilton Anxiety Rating Scale, which has a score range of 0 to 56, where higher scores are associated with higher severity anxiety.
  Score as per below criteria: 0 = Not present, 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Very severe. Total score range of 0-56, where <17 indicates mild severity 18-24 mild to moderate severity 25-30 moderate to severe.
COPE Questionnaire | Screening, day 30, day 60
  Problem-Focused Coping: A high score indicates coping strategies that are aimed at changing the stressful situation. High scores are indicative of psychological strength, grit, a practical approach to problem solving and is predictive of positive outcomes.
  Emotion-Focused Coping: A high score indicates coping strategies that are aiming to regulate emotions associated with the stressful situation. High or low scores are not uniformly associated with psychological health or ill health, but can be used to inform a wider formulation of the respondent's coping styles.
  Avoidant Coping: A high score indicates physical or cognitive efforts to disengage from the stressor. Low scores are typically indicative of adaptive coping.
STAI (State-Trait Anxiety Inventory) | Screening, day 30, day 60
  STAI: State-Trait-Anxiety-Inventory-Score This test consists of 20 items and assesses the current state of anxiety in relation to the current situation in which the patient is to the current situation in which the patient finds herself (State Anxiety) and the general anxiety state existing state of anxiety, which represents a part of her personality (Trait Anxiety).
  The sum score has a range from 20-80. Its interpretation with respective score are discussed below:
  mild anxiety (20 to 39); moderate anxiety (40 to 59); intense anxiety (60 to 80).
visual analogue scale | Screening, day 30, day 60
  Visual analogue scale score- for evaluation of fatigue, nausea, palpitation, breathlessness A higher score (10) represents severe symptoms and a lower score (0) represents no symptoms.
Changes in serum cortisol levels | Screening, day 15, day 60
  The cortisol secretion will be evaluated by measuring morning serum cortisol levels.
Change in serum serotonin levels | Screening, day 30, day 45
  The serotonin secretion will be evaluated by measuring morning serum serotonin levels.
Changes in Modified sleep regularity and medication withdrawal questionnaire (MSRMWQ) | After stopping treatment for 1 week (day 68)
  The Modified Sleep Regularity and Medication Withdrawal Questionnaire (MSRMWQ) is a tool designed to assess changes in sleep patterns and the impact of medication withdrawal on sleep. Total score categories: Part I 00-10 = Poor sleep regularity 21-30 = Better sleep regularity 11-20 = Good sleep regularity 31-40 = Excellent sleep regularity Parameter-wise scoring by 4 point Linkert scale: Part II 0 = No symptom
  1. = Resolved symptom
  2. = Ongoing symptoms requiring no medical assistance
  3. = Ongoing symptoms requiring medical assistance
Change in mood assessed using the Profile of Mood States (POMS) | Screening, day 15, day 30, day 60
  The Profile of Mood States (POMS) is a widely used instrument that measures mood using a 40 item questionnaire with each item rated using a response scale of five categories ranging from "not at all" to "Extremely". Higher score indicates worse mood. Total POMS score categories and stress inference:0-40 = A little; 81-120= Quite a lot; 41-80= Moderately; 121-160= Extremely.

SECONDARY OUTCOMES:
Safety of participant Assessed using adverse events | Screening, baseline, day 15, day 30, day 45, day 60
  It is measure in terms of No. of events
Safety of participant Assessed using treatment compliance and tolerability of investigational product | Screening, baseline, day 15, day 30, day 45, day 60
  It is measure in terms of percentage
Systolic blood pressure difference from reference measurement (mmHg) | Screening, baseline, day 15, day 30, day 45, day 60
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg)
Diastolic blood pressure difference from reference measurement (mmHg) | Screening, baseline, day 15, day 30, day 45, day 60
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg)
Pulse rate difference from reference measurement (beats per minute) | Screening, baseline, day 15, day 30, day 45, day 60
  Assessed against standard clinical grade instrument: Finger-based pulse oximeter (beats per minute)
Complete blood count | Screening and day 60
  White blood cell and platelet count [Thousand per microliter (Thousand/uL)] Red blood cell count [Millions per microliter (million/uL)]
Serum Glutamic Pyruvic Transaminase (SGPT) | Screening and day 60
  Blood level of SGPT was measured. (U/L)
serum glutamic-oxaloacetic transaminase (SGOT) | Screening and day 60
  Blood level of SGOT was measured. (U/L)
Creatinine difference from reference measurement (mg/dl) | Screening and day 60
  Blood levels of Creatinine was measured. (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ramshyam Agarwal, MBBS, DNB, Principal Investigator — Lokmanya Medical Research Centre and Hospital

IPD SHARING:
Plan to Share IPD: No